CLINICAL TRIAL: NCT03306511
Title: Sprint Performance in Football Players With a Previous Hamstring Injury Compared to Healthy Controls: An Exploratory Cross-sectional Study
Brief Title: Sprint Performance in Football Players With a Previous Hamstring Injury
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Lasse Ishøi, MSc, Hvidovre University Hospital
Other Study IDs: SPRINT2017
Record Dates: First submitted 2017-10-05; First posted 2017-10-11 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Sprint Performance; Hamstring Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Football players with a previous self-reported hamstring strain injury in the preceding 12 months
  Interventions: Other: Repeated-sprint test
- Control: Football players without a previous self-reported hamstring strain injury in the preceding 12 months
  Interventions: Other: Repeated-sprint test

INTERVENTIONS:
Other: Repeated-sprint test — 6x30-meter sprint interspersed with 90-s rest

SUMMARY:
Few studies indicate that sprint performance may be impaired in football players with a previous hamstring strain injury. This exploratory cross-sectional study aim to compare sprint performance between football players with and without a previous hamstring strain injury. The findings may elucidate potential indications of insufficient rehabilitation following a hamstring strain injury.

Sprint performance data will be collected using the MySprint Iphone Application.

Due to pragmatic reasons and the exploratory nature of this study the aim is to include players on a team level.

Based on the prevalence of hamstring strain injuries the expected number of cases to be included are 10-20 football players with a previous hamstring strain injury, and a corresponding 80-90 number of healthy controls.

No outcomes will be weighted (flat outcome structure).

ELIGIBILITY:
Inclusion Criteria Controls:

* Able to participate fully in regular football training and matches

Exclusion Criteria Controls:

* Self-reported hamstring strain injury resulting in loss of regular football training sessions or football matches in the preceding 12 months.
* Longstanding injury (>6 weeks) in the lower extremities or trunk in the preceding 12 months.
* Any pain in the lower extremity, pelvis, or spine during testing

Inclusion Criteria Cases:

* Able to participate fully in regular football training and matches
* Self-reported hamstring strain injury resulting in loss of regular football training sessions or football matches in the preceding 12 months.

Exclusion Criteria Cases:

* Longstanding injury (>6 weeks) in the lower extremities (except hamstring strain injury) or trunk in the preceding 12 months.
* Any pain in the lower extremity, pelvis, or spine during testing

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Danish competitive football players
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Theoretical maximal force | Baseline
  Measured using the MySprint Application during a repeated-sprint test consisting of 6x30-m sprints. The outcome measure is exploratory.
Theoretical maximal velocity | Baseline
  Measured using the MySprint Application during a repeated-sprint test consisting of 6x30-m sprints. The outcome measure is exploratory.
Theoritical maximal power output | Baseline
  Measured using the MySprint Application during a repeated-sprint test consisting of 6x30-m sprints. The outcome measure is exploratory.
Slope of the linear decrease on ratio of force as sprint velocity increases | Baseline
  Measured using the MySprint Application during a repeated-sprint test consisting of 6x30-m sprints. The outcome measure is exploratory.

CONTACTS AND LOCATIONS:
Overall Officials: Lasse Ishøi, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Testing will be conducted in the facilities of the included football clubs in Copenhagen, Copenhagen, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided